CLINICAL TRIAL: NCT03124355
Title: Vagal Stimulation in POTS - The Autonomic Inflammatory Reflex (Pilot 3)
Brief Title: Vagal Stimulation in POTS
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Italo Biaggioni, Professor of Medicine and Pharmacology, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 6111
Record Dates: First submitted 2017-04-18; First posted 2017-04-21 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Postural Tachycardia Syndrome
Keywords: vagal stimulation; POTS; galantamine; pyridostigmine
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome | interventions — Pyridostigmine Bromide; Galantamine; Vagus Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, crossover
Who Masked: Participant, Investigator
Masking Description: Participants and investigators will be blinded to the study drugs (placebo, galantamine, pyridostigmine). Participants will be blinded to the vagal stimulation (stimulation vs. sham).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo pill with vagal/sham stimulation (Experimental): Patients will receive a single oral dose of placebo sugar pill, and 1.5-2 hours later they will have two tilt table tests: one with vagal stimulation and one with sham vagal stimulation
  Interventions: Drug: placebo sugar pill; Device: Vagal stimulation; Device: Sham vagal stimulation
- Pyridostigmine with vagal/sham stimulation (Experimental): Patients will receive a single oral dose of pyridostigmine pill 30 mg, and 1.5-2 hours later they will have two tilt table tests: one with vagal stimulation and one with sham vagal stimulation
  Interventions: Drug: Pyridostigmine Pill; Device: Vagal stimulation; Device: Sham vagal stimulation
- Galantamine with vagal/sham stimulation (Experimental): Patients will receive a single oral dose of galantamine pill 8 mg, and 1.5-2 hours later they will have two tilt table tests:one with vagal stimulation and one with sham vagal stimulation
  Interventions: Drug: Galantamine Pill; Device: Vagal stimulation; Device: Sham vagal stimulation

INTERVENTIONS:
Drug: placebo sugar pill — placebo single oral dose
  Other Names: placebo
  Arms: Placebo pill with vagal/sham stimulation
Drug: Pyridostigmine Pill — pyridostigmine bromide 30 mg single oral dose
  Other Names: pyridostigmine bromide; Mestinon
  Arms: Pyridostigmine with vagal/sham stimulation
Drug: Galantamine Pill — Galantamine hydrobromide 8mg single oral dose
  Other Names: Galantamine hydrobromide; Razadyne
  Arms: Galantamine with vagal/sham stimulation
Device: Vagal stimulation — Vagal stimulation will be given at 50 Hz during the tilt table tests
  Other Names: Transcutaneous vagal nerve stimulation
Device: Sham vagal stimulation — Sham vagal stimulation will be given at 0.01 mA during the tilt table tests

SUMMARY:
The purpose of this study is to investigate how the electrical stimulation of a nerve in the skin of the earlobe (transcutaneous vagal nerve stimulation), alone or in combination with two medications (galantamine and pyridostigmine), affects the way the autonomic (involuntary) nervous system controls heart rhythm, symptoms on standing, and inflammatory markers in female patients with postural tachycardia syndrome (POTS). The study consists of 2 parts: a screening (1-2 study days), and 3 testing days. The study will take 5 days total and about 16 participants will be screened for the study. The investigators estimate 13 will be eligible to participate in all of the study days.

DETAILED DESCRIPTION:
This study will test the hypothesis that impairment of the parasympathetic nervous system contributes to the symptoms of POTS and that stimulation of this part of the nervous system improves the excessive increase in heart rate, standing tolerance and inflammation in patients with POTS. For this purpose, the investigators will use electrical stimulation of a nerve in the skin of the earlobe (transcutaneous vagal nerve stimulation) and two medications that increase the levels of acetylcholine (a neurotransmitter) in the central or peripheral nervous system (galantamine and pyridostigmine, respectively) to increase the activity of the parasympathetic nervous system.

Screening Procedures: Potential participants will be screened in the Vanderbilt Autonomic Dysfunction Center (ADC). Medications affecting heart rate, blood pressure, blood volume, inflammatory markers and the autonomic nervous system will be withdrawn for at least five half-lives before studies. Patients will undergo a complete history and physical examination, ECG, routine clinical laboratory analyses and a blood pregnancy test for women of childbearing potential. Autonomic testing including a posture study with plasma catecholamines is then performed to determine if they meet the inclusion/exclusion criteria.

Eligible participants will be studied on three separate days in a randomized, double-blind, crossover fashion. On each testing day, patients will be given one dose of the study medication (either pyridostigmine, galantamine or placebo pill), and then will have two tilt table tests (a motorized table with a footboard that moves to an upright position): one with the vagal stimulation and one with sham electrical stimulation. Heart rhythm, blood pressure and the amount of fluid in the body (body impedance) will be monitored during studies. Blood samples (up to a total of 2 tablespoons per study day) will also be collected. The order of the study days and tilt tests will be decided at random, like the toss of a coin. Each study day will last about 5 hours.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects of 18-45 years, with Postural Tachycardia Syndrome (POTS) as defined by a heart rate increase ≥30 bpm from supine within 10 min of standing or head-up tilt in the absence of orthostatic hypotension, with chronic symptoms (> 6 months), and in the absence of other acute cause of orthostatic tachycardia.
* Subjects able and willing to provide informed consent

Exclusion Criteria:

* Pregnancy.
* Medical conditions that can explain postural tachycardia (e.g., dehydration, medications).
* Patients who are bedridden or chair-ridden
* Subjects taking any medication known to affect autonomic function or inflammatory markers (e.g. corticosteroids) who could not discontinue them before study participation.
* Conditions associated with chronic inflammatory processes which in the investigator's opinion would affect the interpretation of the results. Examples may include smoking, diabetes, BMI>30 kg/m2, current infections or cancer.
* Other factors which in the investigator's opinion would prevent the subject from completing the protocol.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2017-09-30 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
High frequency variability of heart rate | Up to 15 min of head up tilt
  Average of high frequency variability of heart rate during the head up tilt

CONTACTS AND LOCATIONS:
Overall Officials: Italo Biaggioni, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Autonomic Dysfunction Center/ Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No